CLINICAL TRIAL: NCT01268943
Title: Phase 1 Study of Postoperative Capecitabine With Concurrent Radiation in Elderly With Stage II/III Rectal Cancer
Brief Title: Study of Postoperative Concurrent Chemo-radiation With Capecitabine in Elderly Rectal Cancer Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, Jing Jin, M.D., vice chair of radiation department, Chinese Academy of Medical Sciences
Organization: ChineseAMS (Unknown)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CH-GI-013
Record Dates: First submitted 2010-12-28; First posted 2011-01-04 (Estimated); Results first posted 2015-03-17 (Estimated); Last update posted 2015-04-06 (Estimated); Status verified 2015-03

CONDITIONS: Rectal Neoplasms
Keywords: rectal neoplasms; aged; radiotherapy; drug therapy; dose-escalation; capecitabine
MeSH Terms: conditions — Rectal Neoplasms | interventions — Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1000mg (Experimental): capecitabine 1000mg/m2/d d1-14, d22-35 combined with concurrent radiotherapy will be given to enrolled patients.
  Interventions: Drug: Capecitabine
- 1200mg (Experimental): capecitabine 1200mg/m2/d d1-14, d22-35 combined with concurrent radiotherapy will be given to enrolled patients.
  Interventions: Drug: Capecitabine
- 1400mg (Experimental): capecitabine 1400mg/m2/d d1-14, d22-35 combined with concurrent radiotherapy will be given to enrolled patients.
  Interventions: Drug: Capecitabine
- 1500mg (Experimental): capecitabine 1500mg/m2/d d1-14, d22-35 combined with concurrent radiotherapy will be given to enrolled patients.
  Interventions: Drug: Capecitabine

INTERVENTIONS:
Drug: Capecitabine — oral pills, 1000mg/m2/d, split in two times, d1-14, d22-35 combined with concurrent pelvic radiation.
  Other Names: stair 1
  Arms: 1000mg
Drug: Capecitabine — oral pills, 1200mg/m2/d, split in two times, d1-14, d22-35 combined with concurrent pelvic radiation.
  Other Names: stair 2
  Arms: 1200mg
Drug: Capecitabine — oral pills, 1400mg/m2/d, split in two times, d1-14, d22-35 combined with concurrent pelvic radiation.
  Other Names: stair 3
  Arms: 1400mg
Drug: Capecitabine — oral pills, 1500mg/m2/d, split in two times, d1-14, d22-35 combined with concurrent pelvic radiation.
  Other Names: stair 4
  Arms: 1500mg

SUMMARY:
The purpose of this study is to seek the proper dose of capecitabine in post-operative concurrent chemotherapy for stage II/III elderly rectal cancer patients receiving radical surgery, and evaluate the toleration of this modality in such patients.

DETAILED DESCRIPTION:
For those "younger" locally advanced (stage II/III) rectal cancer patients (usually means patients less than 70), it is suggested that after radical surgery, patients should receive concurrent chemo-radiation. Capecitabine is a widely used chemotherapy medicine under such condition. Based on experience, the investigators think this modality can also be tolerated by patients over 70, and will increase local control rate as which has been proved in younger ones. As the first step to test this hypothesis, we designed this phase I study to seek the proper dose of capecitabine, a widely used oral chemotherapy medicine, in postoperative concurrent chemo-radiation for stage II/III rectal cancer patients over 70, and to evaluate the safety of this modality in this group of patients.

ELIGIBILITY:
Inclusion Criteria:

* rectal adenocarcinoma, pathological stage II/III(T3-4 or N+, UICC 2002), radical surgery received.
* interval between surgery and enrollment no less than two week and no more than 3 months.
* KPS status no less than 70; life expectancy no less than 6 months.
* without life-threatening complications, such as severe hypertension, coronary heart disease, cerebral vascular disease, uncontrolled diabetes, etc.
* without severe drug allergy history.
* hemoglobin >= 100g/L, white blood cell >= 3.5*10E9/L, neutrophil >= 1.5*10E9/L, platelet >= 100*10E9/L.
* Creatin <= 1.5* ULN(upper limit of normal), Total bilirubin <= 2.5 ULN, AST and AST <= 2.5* ULN, AKP <= 2.5*ULN
* do not receive chemotherapy before six months from enrollment.
* no previously pelvic irradiation history
* informed consent signed

Exclusion Criteria:

* other cancer history, except curable non-melanoma skin cancer or cervix in-situ carcinoma
* allergy history to thymidine phosphorylase
* previous pelvic irradiation history
* receiving adjuvant chemotherapy in six months before enrollment
* active infection existed
* severe complication, such as acute myocardial infarction in 6 months, uncontrolled diabetes ( Plasma glucose concentrations in any time of a day≥11.1mmol/L）, severe cardiac arrhythmia， etc.
* life expectancy less than 6 months
* estimated cannot finish treatment
* attend other clinical trials in four weeks before enrollment
* receive other anti-cancer treatment currently
* other conditions which regarded illegal by censors with full reasons. for example, some conditions may conflict from the protocol.

Min Age: 71 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 18 (Actual)
Dates: Start 2010-11; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jing Jin, Ph.D., Principal Investigator — radiation department, cancer hospital, CAMS; Yexiong Li, Ph.D., Principal Investigator — Radiation Department, Cancer Hospital, CAMS
Locations (1):
- radiation department, Cancer Hospital, CAMS, Beijing, Beijing Municipality, China

REFERENCES:
- [Background] Colorectal Cancer Collaborative Group. Adjuvant radiotherapy for rectal cancer: a systematic overview of 8,507 patients from 22 randomised trials. Lancet. 2001 Oct 20;358(9290):1291-304. doi: 10.1016/S0140-6736(01)06409-1. PMID 11684209
- [Background] Tveit KM, Guldvog I, Hagen S, Trondsen E, Harbitz T, Nygaard K, Nilsen JB, Wist E, Hannisdal E. Randomized controlled trial of postoperative radiotherapy and short-term time-scheduled 5-fluorouracil against surgery alone in the treatment of Dukes B and C rectal cancer. Norwegian Adjuvant Rectal Cancer Project Group. Br J Surg. 1997 Aug;84(8):1130-5. PMID 9278661
- [Background] Fisher B, Wolmark N, Rockette H, Redmond C, Deutsch M, Wickerham DL, Fisher ER, Caplan R, Jones J, Lerner H, et al. Postoperative adjuvant chemotherapy or radiation therapy for rectal cancer: results from NSABP protocol R-01. J Natl Cancer Inst. 1988 Mar 2;80(1):21-9. doi: 10.1093/jnci/80.1.21. PMID 3276900
- [Background] Krook JE, Moertel CG, Gunderson LL, Wieand HS, Collins RT, Beart RW, Kubista TP, Poon MA, Meyers WC, Mailliard JA, et al. Effective surgical adjuvant therapy for high-risk rectal carcinoma. N Engl J Med. 1991 Mar 14;324(11):709-15. doi: 10.1056/NEJM199103143241101. PMID 1997835
- [Background] Wolmark N, Wieand HS, Hyams DM, Colangelo L, Dimitrov NV, Romond EH, Wexler M, Prager D, Cruz AB Jr, Gordon PH, Petrelli NJ, Deutsch M, Mamounas E, Wickerham DL, Fisher ER, Rockette H, Fisher B. Randomized trial of postoperative adjuvant chemotherapy with or without radiotherapy for carcinoma of the rectum: National Surgical Adjuvant Breast and Bowel Project Protocol R-02. J Natl Cancer Inst. 2000 Mar 1;92(5):388-96. doi: 10.1093/jnci/92.5.388. PMID 10699069
- [Background] Gastrointestinal Tumor Study Group. Prolongation of the disease-free interval in surgically treated rectal carcinoma. N Engl J Med. 1985 Jun 6;312(23):1465-72. doi: 10.1056/NEJM198506063122301. PMID 2859523
- [Background] Hoff PM, Ansari R, Batist G, Cox J, Kocha W, Kuperminc M, Maroun J, Walde D, Weaver C, Harrison E, Burger HU, Osterwalder B, Wong AO, Wong R. Comparison of oral capecitabine versus intravenous fluorouracil plus leucovorin as first-line treatment in 605 patients with metastatic colorectal cancer: results of a randomized phase III study. J Clin Oncol. 2001 Apr 15;19(8):2282-92. doi: 10.1200/JCO.2001.19.8.2282. PMID 11304782
- [Background] Van Cutsem E, Twelves C, Cassidy J, Allman D, Bajetta E, Boyer M, Bugat R, Findlay M, Frings S, Jahn M, McKendrick J, Osterwalder B, Perez-Manga G, Rosso R, Rougier P, Schmiegel WH, Seitz JF, Thompson P, Vieitez JM, Weitzel C, Harper P; Xeloda Colorectal Cancer Study Group. Oral capecitabine compared with intravenous fluorouracil plus leucovorin in patients with metastatic colorectal cancer: results of a large phase III study. J Clin Oncol. 2001 Nov 1;19(21):4097-106. doi: 10.1200/JCO.2001.19.21.4097. PMID 11689577
- [Background] Van Cutsem E, Hoff PM, Harper P, Bukowski RM, Cunningham D, Dufour P, Graeven U, Lokich J, Madajewicz S, Maroun JA, Marshall JL, Mitchell EP, Perez-Manga G, Rougier P, Schmiegel W, Schoelmerich J, Sobrero A, Schilsky RL. Oral capecitabine vs intravenous 5-fluorouracil and leucovorin: integrated efficacy data and novel analyses from two large, randomised, phase III trials. Br J Cancer. 2004 Mar 22;90(6):1190-7. doi: 10.1038/sj.bjc.6601676. PMID 15026800
- [Background] Zhu AX, Willett CG. Chemotherapeutic and biologic agents as radiosensitizers in rectal cancer. Semin Radiat Oncol. 2003 Oct;13(4):454-68. doi: 10.1016/S1053-4296(03)00048-1. PMID 14586834
- [Background] Souglakos J, Androulakis N, Mavroudis D, Kourousis C, Kakolyris S, Vardakis N, Kalbakis K, Pallis A, Ardavanis A, Varveris C, Georgoulias V. Multicenter dose-finding study of concurrent capecitabine and radiotherapy as adjuvant treatment for operable rectal cancer. Int J Radiat Oncol Biol Phys. 2003 Aug 1;56(5):1284-7. doi: 10.1016/s0360-3016(03)00275-x. PMID 12873672
- [Background] Dunst J, Reese T, Sutter T, Zuhlke H, Hinke A, Kolling-Schlebusch K, Frings S. Phase I trial evaluating the concurrent combination of radiotherapy and capecitabine in rectal cancer. J Clin Oncol. 2002 Oct 1;20(19):3983-91. doi: 10.1200/JCO.2002.02.049. PMID 12351595
- [Background] Ngan SY, Michael M, Mackay J, McKendrick J, Leong T, Lim Joon D, Zalcberg JR. A phase I trial of preoperative radiotherapy and capecitabine for locally advanced, potentially resectable rectal cancer. Br J Cancer. 2004 Sep 13;91(6):1019-24. doi: 10.1038/sj.bjc.6602106. PMID 15305186
- [Background] Aapro MS, Kohne CH, Cohen HJ, Extermann M. Never too old? Age should not be a barrier to enrollment in cancer clinical trials. Oncologist. 2005 Mar;10(3):198-204. doi: 10.1634/theoncologist.10-3-198. PMID 15793223
- [Background] Folprecht G, Cunningham D, Ross P, Glimelius B, Di Costanzo F, Wils J, Scheithauer W, Rougier P, Aranda E, Hecker H, Kohne CH. Efficacy of 5-fluorouracil-based chemotherapy in elderly patients with metastatic colorectal cancer: a pooled analysis of clinical trials. Ann Oncol. 2004 Sep;15(9):1330-8. doi: 10.1093/annonc/mdh344. PMID 15319237
- [Background] Jin J, Li YX, Liu YP, Wang WH, Song YW, Li T, Li N, Yu ZH, Liu XF. A phase I study of concurrent radiotherapy and capecitabine as adjuvant treatment for operable rectal cancer. Int J Radiat Oncol Biol Phys. 2006 Mar 1;64(3):725-9. doi: 10.1016/j.ijrobp.2005.08.017. Epub 2005 Oct 19. PMID 16242260
- [Background] Abir F, Alva S, Longo WE. The management of rectal cancer in the elderly. Surg Oncol. 2004 Dec;13(4):223-34. doi: 10.1016/j.suronc.2004.08.008. PMID 15615660
- [Background] Pasetto LM, Monfardini S. The role of capecitabine in the treatment of colorectal cancer in the elderly. Anticancer Res. 2006 May-Jun;26(3B):2381-6. PMID 16821620
- [Background] Dobie SA, Warren JL, Matthews B, Schwartz D, Baldwin LM, Billingsley K. Survival benefits and trends in use of adjuvant therapy among elderly stage II and III rectal cancer patients in the general population. Cancer. 2008 Feb 15;112(4):789-99. doi: 10.1002/cncr.23244. PMID 18189291
- [Background] Papamichael D, Audisio R, Horiot JC, Glimelius B, Sastre J, Mitry E, Van Cutsem E, Gosney M, Kohne CH, Aapro M; SIOG. Treatment of the elderly colorectal cancer patient: SIOG expert recommendations. Ann Oncol. 2009 Jan;20(1):5-16. doi: 10.1093/annonc/mdn532. Epub 2008 Oct 15. PMID 18922882
- [Background] Fiorica F, Cartei F, Carau B, Berretta S, Sparta D, Tirelli U, Santangelo A, Maugeri D, Luca S, Leotta C, Sorace R, Berretta M. Adjuvant radiotherapy on older and oldest elderly rectal cancer patients. Arch Gerontol Geriatr. 2009 Jul-Aug;49(1):54-9. doi: 10.1016/j.archger.2008.05.001. Epub 2008 Jun 24. PMID 18573548
- [Background] Surgery for colorectal cancer in elderly patients: a systematic review. Colorectal Cancer Collaborative Group. Lancet. 2000 Sep 16;356(9234):968-74. PMID 11041397
- [Background] Potosky AL, Harlan LC, Kaplan RS, Johnson KA, Lynch CF. Age, sex, and racial differences in the use of standard adjuvant therapy for colorectal cancer. J Clin Oncol. 2002 Mar 1;20(5):1192-202. doi: 10.1200/JCO.2002.20.5.1192. PMID 11870160
- [Background] Bouvier AM, Launoy G, Lepage C, Faivre J. Trends in the management and survival of digestive tract cancers among patients aged over 80 years. Aliment Pharmacol Ther. 2005 Aug 1;22(3):233-41. doi: 10.1111/j.1365-2036.2005.02559.x. PMID 16091061
- [Background] Goldberg RM, Tabah-Fisch I, Bleiberg H, de Gramont A, Tournigand C, Andre T, Rothenberg ML, Green E, Sargent DJ. Pooled analysis of safety and efficacy of oxaliplatin plus fluorouracil/leucovorin administered bimonthly in elderly patients with colorectal cancer. J Clin Oncol. 2006 Sep 1;24(25):4085-91. doi: 10.1200/JCO.2006.06.9039. PMID 16943526
- [Background] Feliu J, Sereno M, Castro JD, Belda C, Casado E, Gonzalez-Baron M. Chemotherapy for colorectal cancer in the elderly: Whom to treat and what to use. Cancer Treat Rev. 2009 May;35(3):246-54. doi: 10.1016/j.ctrv.2008.11.004. Epub 2009 Apr 2. PMID 19345021

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between October 2010 and November 2013, 18 patients were enrolled in a hospital.
Period: Overall Study
Arm/Group | 1000mg | 1200mg | 1400mg | 1500mg
Started | 6 | 3 | 3 | 6
Completed | 6 | 3 | 3 | 6
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- 1000mg: capecitabine 500mg/m2 twice daily. 6 patients enrolled
- 1200mg: capecitabine 600mg/m2 twice daily. 3 patients enrolled
- 1400mg: capecitabine 700mg/m2 twice daily. 3 patients enrolled
- 1500mg: capecitabine 750mg/m2 twice daily. 6 patients enrolled
- Total: Total of all reporting groups
Arm/Group | 1000mg | 1200mg | 1400mg | 1500mg | Total
Number analyzed (Participants) | 6 | 3 | 3 | 6 | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0 | 0 | 0
  >=65 years | 6 | 3 | 3 | 6 | 18
Age, Continuous [Mean (Full Range); unit: years] | 75.5 [72 to 83] | 73.7 [73 to 75] | 75.7 [71 to 81] | 73.5 [70 to 78] | 74.5 [70 to 83]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 0 | 4 | 5
  Male | 5 | 3 | 3 | 2 | 13

OUTCOME MEASURES:

1. Primary Outcome: Dose Related Toxicity
Description: dose related toxicity is defined as follows:1. WBC damage >= grade 3; granular cell decrease >= grade 3; hemoglobin >= grade 2; platelet >= grade 2;SGPT/SGOT elevation >= grade 2; ALP >= grade 2; GGT >= grade 2; Tbil >= grade 2;renal function damage: BUN/Cr elevation >= grade 2;Non-gradular cell decreased fever >= grade 2;nausea/vomiting >= grade 2; fatigue >= grade 3; weight loss >= grade 3;gastritis >= grade 3; dairrea >= grade 3; abdominal pain >= grade 3; pancreatitis >= grade 2; upper gastrointestinal bleeding >= grade 2;other toxic reaction >= grade 3;KPS < 50 during the treatment
Time Frame: up to 9 weeks
Measure: Number; unit: event
Arm/Group | 1000mg | 1200mg | 1400mg | 1500mg
Number analyzed (Participants) | 6 | 3 | 3 | 6
event | 1 | 0 | 0 | 3

ADVERSE EVENTS:
Time Frame: 9 weeks
Arm/Group | 1000mg | 1200mg | 1400mg | 1500mg
Serious Adverse Events (participants affected / at risk) | 1/6 | 0/3 | 0/3 | 2/6
Other Adverse Events (participants affected / at risk) | 5/6 | 2/3 | 3/3 | 5/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1000mg (N=6) | 1200mg (N=3) | 1400mg (N=3) | 1500mg (N=6)
Diarrhea, grade 3 (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
vomiting, grade 3 (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
leukopenia, grade 3 (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1000mg (N=6) | 1200mg (N=3) | 1400mg (N=3) | 1500mg (N=6)
fatigue (General disorders) | 4 (4) | 2 (2) | 2 (2) | 3 (3)
anorexia (General disorders) | 3 (3) | 2 (2) | 2 (2) | 3 (3)
vomiting, grade 1-2 (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
diarrhea, grade 1-2 (Gastrointestinal disorders) | 3 (3) | 0 (0) | 1 (1) | 2 (2)
incontinence (Gastrointestinal disorders) | 3 (3) | 1 (1) | 0 (0) | 1 (1)
abodminal pain (Gastrointestinal disorders) | 3 (3) | 1 (1) | 0 (0) | 1 (1)
skin reation (Skin and subcutaneous tissue disorders) | 4 (4) | 2 (2) | 2 (2) | 2 (2)
hand-foot syndrome (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
leukopenia, grade 1-2 (Blood and lymphatic system disorders) | 5 (5) | 2 (2) | 2 (2) | 4 (4)
thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No